CLINICAL TRIAL: NCT05836168
Title: Effects of Microbiome Modulation on Sleep in Working People: A Randomized Controlled Pilot Trial
Brief Title: Effects of Microbiome Modulation on Sleep in Working People
Acronym: Sleep
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: CBmed Ges.m.b.H. (Other)
Responsible Party: Principal Investigator, Vanessa Stadlbauer-Koellner, MD, Univ. Prof. PD Dr. med, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 35-176 ex 22/23
Record Dates: First submitted 2023-04-18; First posted 2023-05-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: placebo, outcome assessors are blinded to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): multi-strain probiotic mixture containing Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Bifidobacterium lactis W52, Lactobacillus acidophilus W22, Lactobacillus casei W56, Lactobacillus paracasei W20, Lactobacillus plantarum W62, Lactobacillus salivarius W24, Lactococcus lactis W19 in a matrix of maize starch, maltodextrin, inulin, potassium chloride, rice protein, magnesium sulfate, fructooligosaccharides, amylases and mangane sulfate at a dose of 2 x 3g per day for 4 weeks.
  Interventions: Dietary Supplement: Omnibiotic Stress Repair
- Placebo (Placebo Comparator): 2 x 3g of a similar looking and tasting placebo per day for 4 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omnibiotic Stress Repair — multispecies probiotic
  Other Names: Omnibiotic Stress
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
We aim to test whether quality of sleep in working people can be improved by modulating the gut microbiome with probiotics.

DETAILED DESCRIPTION:
A good night´s sleep is essential for our attention, cognition and mood. Sleep fragmentation can therefore lead to poor performance, loss of productivity, and errors, incidents and accidents in the workplace. Sleep disruption has further been associated with metabolic and cardiovascular diseases, psychiatric diseases and cancer.The gut microbiome and its metabolites exhibit diurnal rhythmicity in response to food intake and influence human clock gene expression and sleep duration. Sleep fragmentation causes dysbiosis and hormonal disturbances. First data from animal experiments and small human studies imply that modulation of the gut microbiome may improve sleep quality and thereby mental and physical health. Probiotics can alter the gut microbiota composition and can mitigate positive effects on psychiatric symptoms via the microbiome gut-brain axis by metabolites such as short-chain fatty acids (SCFA) that can pass the blood-brain barrier and thereby comprise a potential strategy to improve sleep quality and other quality of life related outcomes. Evidence on the effect of probiotics to improve quality of sleep is available from several small-scale clinical studies in different populations. The benefit seems to be stronger in people under physical or mental stress.

Also, a large marketing survey conducted in Germany in over >10.000 consumers indicated that a multispecies probiotic, that has been described to improve inflammation, gut barrier dysfunction and immune function in different patient cohorts is able to improve sleep quality and quality of life, however since this study was non-randomized, a bias cannot be excluded.

Understanding the interaction between the gut microbiome, chronobiology and health is therefore of high importance and in line with the United Nations' Sustainable Development Goal 3 of the 2030 Agenda for Sustainable Development to "ensure healthy lives and promoting well-being for all at all ages".

ELIGIBILITY:
Inclusion criteria

* Age >18
* Working
* Signed Informed Consent;
* Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data for at least 15 years
* Pittsburgh Sleep Quality index score of >5 Exclusion criteria
* Diagnosed with a gastrointestinal infection within 4 weeks prior to screening
* Severe gastrointestinal diseases (e.g. inflammatory bowel diseases)
* Received any of the following products/medication within 4 weeks prior to screening: systemic antibiotics, prokinetics, prebiotic supplements, probiotic supplements
* Concomitant diseases or other circumstances that suggest that the patients are not eligible for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in subjective sleep quality | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
sleep latency | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)
sleep duration | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)
habitual sleep efficiency | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)
sleep disturbances | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)
use of sleeping medication | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)
daytime dysfunction | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Quality of life | 4 weeks
  short form 12 (SF-12)
perceived stress levels | 4 weeks
  measured by perceived stress questionnaire (PSQ-20)
Gastrointestinal quality of life | 4 weeks
  measured by gastrointestinal quality of life index (GIQLI)

OTHER OUTCOMES:
Microbiome composition | 4 weeks
  16s rDNA analysis, beta diversity
Metabolite composition | 4 weeks
  NMR metabolomics
Hair Cortisol levels | 4 weeks
  Hair cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided
Depending on the results, according to the grant contract, IPR will be shared among partners and after these discussions IPD may be shared. Microbiome sequencing data will be deposited in a public repository